CLINICAL TRIAL: NCT03844867
Title: ALMOND1: Nutritional, Organoleptic and Motility Profile of Toritto & Californian Almond
Brief Title: Healthy Properties of Two Almond Varieties. CEA vs. CARMEL
Acronym: ALMOND1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, piero portincasa, Professor, University of Bari
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 5037
Record Dates: First submitted 2019-02-11; First posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Filippo Cea and Carmel (Experimental): Subjects <65 years.
  Interventions: Dietary Supplement: Filippo Cea and Carmel

INTERVENTIONS:
Dietary Supplement: Filippo Cea and Carmel — Subjects will be given a subjective organoleptic assessment of both the almonds (Filippo Cea and Carmel) administered blindly and randomly.
  Motility test: Each subject will be subjected to gastrointestinal motility study according to international guidelines, i.e. he will be evaluated in 3 different days. The test will be made in response to test-meal ('NutriDrink') or Filippo Cea almonds (12 gr. fat=24 gr. almonds) or Carmel almonds (12 gr. fat = 24 gr. almonds).

SUMMARY:
The cultivation of almond (Amygdalus communis L.) has always been a hallmark of the Mediterranean, representing a resource both food and economic. Almonds are high in fat (55.3%, mainly (39.4%) they consist of MUFA), are an excellent source of vitamin E, manganese, magnesium, copper, phosphorus, fiber, riboflavin and protein, phenolic and polyphenolic.

Numerous studies correlate moderate and regular consumption of nuts with an important role in health. In particular, habitual almond consumption does not lead to weight gain, and their inclusion in low-calorie diets appears to promote more weight loss than a comparable carbohydrate-based low-calorie diet. Also, almonds have a low glycemic index and do not adversely impact insulin sensitivity. So they reduce certain risk factors linked to diabetes and cardiovascular disease. Almonds are an excellent source of bioavailable α-tocopherol, and increasing their intake enhances the resistance of LDL against oxidation. In addition, the polyphenolic constituents of almonds have been characterized recently and found to possess antioxidant actions. Some studies show as consumption of almonds has been shown to be associated with lower levels of serum cholesterol and triglycerides thanks of their poly-unsaturated fatty acids.

Despite Mediterranean countries have dominated world trade for a long time, from the '80 years, Italy underwent a strong production crisis, mainly due to the lack of new plants conducted according to the most modern techniques of cultivation and competition from other crops considered more profitable (e.g. wine, horticultural and citrus). The United States, in particular California, currently control more than a third of the world production of almond, using different cultivars and agronomic practices, based on more modern systems.

In Apulia, various native cultivars have been developed such as "Filippo Cea", which have resisted the invasion of the most productive varieties of California.

The aim of the project is to assess the quality and the beneficial effects of almonds, comparing a local cultivar (Filippo Cea) with an imported (Carmel) one. The study will be characterized by different phases:

* Organoleptic analysis of the two different cultivars of almonds
* evaluation of gastrointestinal motility after taking the two types of almonds.

DETAILED DESCRIPTION:
The cultivation of almond (Amygdalus communis L.) has always been a hallmark of the Mediterranean, representing a resource both food and economic. To traditional uses, mostly related the confectionery industry, they are added other in cosmetics.

The plant is perfectly adapted to the Mediterranean climate, characterized by hot, dry summers, and is often associated to olive, carob and fig trees, species with similar climatic requirements. Almonds are a nutrient-dense food. They are high in fat (55.3%), mainly (39.4%) they consist of monounsaturated fatty acids (MUFA). Moreover, almonds are an excellent source of vitamin E, manganese, magnesium, copper, phosphorus, fibre, riboflavin and protein. In addition, almond proteins are unusually high in arginine and possess good digestibility. Recent studies have shown that almonds also contain a diverse array of phenolic and polyphenolic.

Numerous studies correlate the moderate and regular consumption of nuts with an important role in health. In particular, habitual almond consumption does not lead to weight gain, and their inclusion in low-calorie diets appears to promote more weight loss than a comparable carbohydrate-based low-calorie diet. Also, almonds have a low glycemic index and do not adversely impact insulin sensitivity. So they reduce certain risk factors linked to diabetes and cardiovascular disease. Almonds are an excellent source of bioavailable α-tocopherol, and increasing their intake enhances the resistance of LDL against oxidation. In addition, the polyphenolic constituents of almonds have been characterized recently and found to possess antioxidant actions. Some studies show as consumption of almonds has been shown to be associated with lower levels of serum cholesterol and triglycerides thanks of their polyunsaturated fatty acids.

They are also indicated in the diet of elderly people by helping to increase bone mineral density. Important is also the antibacterial and antifungal power of almond oils shown in recent years.

Despite Mediterranean countries (particularly Spain and Italy) have dominated world trade for a long time, from the '80 years, Italy underwent a strong production crisis, mainly due to the lack of new plants conducted according to the most modern techniques of cultivation and competition from other crops considered more profitable (eg. wine, horticultural and citrus). The United States currently control more than a third of the world production of almond, using different cultivars and agronomic practices, based on more modern systems. Californian industry is characterized by much larger companies than Italian and modern mechanized harvesting systems linked to the condition of serious shortage of manpower. This allowed it to create a standardized product with no impurities, selected and beautifully packaged who conquered large segments of trade, while not offering a high standard from the point of view of the qualitative composition.

In Apulia, almond of Toritto has spread on the border between pre-Murgia and Alta Murgia which takes its name from the country where it is produced. Here various native cultivars have been developed such as "Filippo Cea", the "Antonio De Vito" and "Genco", which have resisted the invasion of the most productive varieties of California. Almond of Toritto is a product of excellence, recognized as typical Apulian product, entered in the list of Italian traditional food products of the Ministry of Agriculture, Food and Forestry.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers.
* Aged 18-80 years old.
* Normal and obese subjects.
* Able to provide informed consent.

Exclusion Criteria:

* Refusal to sign the informed consent.
* Diagnosis of organic diseases including neoplastic inflammatory illness or cardiovascular diseases.
* Hypersensibility to almonds.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Organoleptic valuations | 1 day
  Subjects will give a subjective organoleptic assessment of both the almonds (Filippo Cea and Carmel) administered blindly and randomly. A semiquantitative scale (ranging from 0 to 3, in order of ascertainment for sensations, from lower=0 to higher=3 grade) will be used as markers of visual aspects, olfactory, flavor, mouth tactile sensations. Before each test, and also between the two samples, the mouth will be washed with mineral water. Food, drink, smoking and physical activity will not be allowed before and during the test.
Visual Analog Scale | 1 day
  A quantitative visual analogue scale (VAS, ranging from 0 to 100 mm on a horizontal line, from lower to higher ascertainment for sensations) will be used as markers of visual aspects, olfactory, flavor, mouth tactile sensations.
Ultrasound examination (gallbladder, stomach) and orocecal transit time) | 3 days
  Each subject will be subjected to gastrointestinal motility study according to international guidelines, i.e. he will be evaluated in 3 different days, in the morning in the fasting state to monitor gastric empting, gallbladder empting (ultrasound) and oro-cecal transit time (H 2 lactulose BT), at baseline and at 5 minutes intervals during the firsts 30 minutes, and at 15 minutes intervals during the remaining 90 minutes, for a total of 2 hours of observations. The test will be made in response to test-meal ('NutriDrink') or Filippo Cea almonds (12 gr. fat=24 gr. almonds) or Carmel almonds (12 gr. fat = 24 gr. almonds).

CONTACTS AND LOCATIONS:
Overall Officials: Piero Portincasa, MD, PhD, Principal Investigator — Department of Biomedical Sciences and Human Oncology - Clinica Medica "A. Murri"
Locations (1):
- Department of Biomedical Sciences and Human Oncology - Clinica medica "A. Murri", Bari, BA, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ahrens S, Venkatachalam M, Mistry AM, Lapsley K, Sathe SK. Almond (Prunus dulcis L.) protein quality. Plant Foods Hum Nutr. 2005 Sep;60(3):123-8. doi: 10.1007/s11130-005-6840-2. PMID 16187015
- [Background] Wu X, Beecher GR, Holden JM, Haytowitz DB, Gebhardt SE, Prior RL. Lipophilic and hydrophilic antioxidant capacities of common foods in the United States. J Agric Food Chem. 2004 Jun 16;52(12):4026-37. doi: 10.1021/jf049696w. PMID 15186133
- [Background] Jenkins DJ, Kendall CW, Marchie A, Parker TL, Connelly PW, Qian W, Haight JS, Faulkner D, Vidgen E, Lapsley KG, Spiller GA. Dose response of almonds on coronary heart disease risk factors: blood lipids, oxidized low-density lipoproteins, lipoprotein(a), homocysteine, and pulmonary nitric oxide: a randomized, controlled, crossover trial. Circulation. 2002 Sep 10;106(11):1327-32. doi: 10.1161/01.cir.0000028421.91733.20. PMID 12221048